CLINICAL TRIAL: NCT05003401
Title: Leveraging Technological Advancements to Improve the Treatment of Trichotillomania
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00279950
Record Dates: First submitted 2021-08-06; First posted 2021-08-12 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Trichotillomania (Hair-Pulling Disorder); Trichotillomania; Hair Pulling
MeSH Terms: conditions — Trichotillomania

STUDY DESIGN:
Intervention Model Description: Participants will be provided with the Keen2 wrist-worn device to determine whether this device increases awareness of automatic hair pulling behaviors over a period of 4 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HabitAware Keen 2 (Experimental): Participants will receive the wrist device device that alerts the participant when the participant is engaging in hair pulling behavior.
  Interventions: Device: HabitAware Keen2

INTERVENTIONS:
Device: HabitAware Keen2 — Participants will receive an awareness bracelet to be worn on the dominant wrist over a period of 4 weeks. The bracelet device will vibrate when the participant is engaging in hair pulling behaviors. As hair pulling behaviors may occur outside of awareness (i.e., automatic pulling behaviors), this vibration and detection is anticipated to increase the participants awareness of hair pulling behaviors.

SUMMARY:
This project will examine the effect using the Keen 2 on hair pulling styles (automatic and focused), the severity of hair pulling behaviors, and related psychiatric symptoms. Given that the Keen2 is anticipated to increase awareness of pulling behavior (but not necessarily change pulling behavior), the investigators hypothesize that the Keen 2 will increase awareness of pulling behaviors and reduce automatic pulling behavior. The investigators will explore reductions in overall hair pulling severity and related psychiatric symptoms.

DETAILED DESCRIPTION:
Novel technologies present one solution to help identify and reduce automatic pulling behaviors associated with trichotillomania (TTM). The Keen 2 is one such novel technology, which is a bracelet which gives the user alerts in the form of a vibration when the user is engaging in hair pulling behavior. Thus, using the Keen 2 could positively increase the awareness of automatic pulling behaviors, which is largely unaffected by existing evidence-based treatments like HRT. This information would be advantageous for the scientific community to determine the possible benefit of this approach to help individuals with TTM.

This project will examine the effect using the Keen 2 on hair pulling styles (automatic and focused), the severity of hair pulling behaviors, and related psychiatric symptoms. Given that the Keen2 is anticipated to increase awareness of pulling behavior (but not necessarily change pulling behavior), the investigators hypothesize that the Keen 2 will increase awareness of pulling behaviors and reduce automatic pulling behavior. The investigators will explore reductions in overall hair pulling severity and related psychiatric symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older;
2. meet diagnostic criteria for TTM using the TDI-R
3. have a MGH-HPS total score ≥ 12 at baseline;

(3) have an "automatic" pulling score ≥ 15 on the MIST; (4) able to wear the Keen2 device for four weeks; (5) able to attend three study visits; (6) unmedicated or a stable dose of psychiatric medication for 8 weeks prior to enrollment; (7) be English speaking.

Exclusion Criteria:

1. an inability to complete rating scales, and
2. an inability to attend study visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-11-17 (Actual); Primary Completion 2024-07-16 (Actual); Study Completion 2024-07-16 (Actual)

PRIMARY OUTCOMES:
Milwaukee Inventory for Subtypes of Trichotillomania-Adult Version | 1 week
  The Milwaukee Inventory for Subtypes of Trichotillomania-Adult Version (MIST-A) is a 15-item self-report measure that assesses automatic (5-items) and focused (10-items) hair-pulling styles. Items are rated on a 10-point Likert scale from 0=not true of any of my hair pulling to 9= true for all of my hair pulling. Items are summed to produce an automatic hair pulling (range: 0 - 45) and focused hair pulling score (range: 0 - 90). Higher scores suggest greater presence of this hair pulling behavior. The MIST-A has demonstrated good reliability and validity.

SECONDARY OUTCOMES:
Massachusetts General Hospital Hair Pulling Scale | 1 week
  The Massachusetts General Hospital Hair Pulling Scale (MGH-HPS) is a 7-item self-report measure assessing urges to pull, actual pulling, perceived control, and associated distress. The items are rated on a 5-point Likert scale ranging from 0 to 4, with a total score derived from the summation of all 7-items (range: 0 to 28). Higher total scores are indicative of greater hair pulling severity. The MGH-HPS exhibited good internal consistency with strong test-retest reliability between 2 and 4 weeks. Convergent validity for the MGH-HPS received support from significant correlations within measurement type. Discriminant validity was demonstrated by non-significant correlations with ratings of depression. The MGH-HPS has been used as a treatment outcome measure and appears to be sensitive to behavioral and pharmacological treatments in a sample that included both youth and adults (McGuire et al., 2012).

CONTACTS AND LOCATIONS:
Overall Officials: Joseph McGuire, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No